CLINICAL TRIAL: NCT05514873
Title: A Phase 3b, Multicenter, Open-Label, Single-Arm Study to Evaluate the Safety, Tolerability, and Efficacy of Zilucoplan in Participants With Generalized Myasthenia Gravis Switching From Intravenous Complement Component 5 Inhibitors to Subcutaneous Zilucoplan
Brief Title: An Open-label Study to Evaluate the Safety, Tolerability, and Efficacy of Subcutaneous Zilucoplan in Participants With Generalized Myasthenia Gravis Who Were Previously Receiving Intravenous Complement Component 5 Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0017
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Generalized Myasthenia Gravis
Keywords: gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.3 mg/kg zilucoplan (RA101495) (Experimental): Study participants will be treated with subcutaneous zilucoplan (0.3mg/kg/day)
  Interventions: Drug: zilucoplan (RA101495)

INTERVENTIONS:
Drug: zilucoplan (RA101495) — Subcutaneous injection

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of switching from intravenous (IV) complement component 5 (C5) inhibitors to subcutaneous (SC) Zilucoplan in study participants with generalized myasthenia gravis (gMG)

ELIGIBILITY:
Inclusion Criteria:

* Participant has been treated with an intravenous (IV) complement component 5 (C5) inhibitor approved for the treatment of generalized myasthenia gravis (gMG) at the recommended dose regimen for at least 3 months (for eculizumab) or 4 months (for ravulizumab) prior to Screening with a clinically stable disease as per the Investigator's judgment.
* Participant is willing to switch from his/her current IV C5 inhibitor to subcutaneous (SC) zilucoplan (ZLP)
* Participant has a documented diagnosis of gMG (Myasthenia Gravis Foundation of America; MGFA Class II-IVa) at Screening based on participant history and supported by previous evaluations
* Participant has a well-documented record of positive serology for acetylcholine receptor binding autoantibodies prior to Screening
* Participant has no more than a 2-point change in Myasthenia Gravis-Activities of Daily Living (MG-ADL) score at Baseline compared with the Screening Visit
* Participant has had no change in corticosteroid dose during the Screening Period and no change in corticosteroid dose is anticipated to occur during the 12-week Main Treatment Period
* Participant has had no change in immunosuppressive therapy, including dose, during the Screening Period and no change in immunosuppressive therapy is anticipated to occur during the 12-week Main Treatment Period
* Participant has a record of vaccination with at least 1 dose of a quadrivalent meningococcal vaccine and meningococcal serotype B vaccine at least 14 days prior to the first dose of ZLP if not vaccinated within 3 years prior to the start of study medication
* Male and/or female
* A male participant is recommended to agree to use contraception during the study and for at least 40 days (5 half lives) after the last dose of study medication, and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant; not breastfeeding, and at least one of the following conditions applies:
* Not a woman of childbearing potential (WOCBP) OR
* A WOCBP who agrees to follow the contraceptive guidance during the study and for at least 40 days (5 half lives) after the last dose of study medication.
* Participant is capable of giving signed informed consent

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the participant's ability to participate in this study
* Participant has a known hypersensitivity to any components of the study medication as stated in this protocol
* Participant has had a thymectomy within 6 months prior to Baseline or has one scheduled to occur during the 12-week Main Treatment Period
* Participant has a history of meningococcal disease
* Participant has or has had a current or recent systemic infection within 2 weeks prior to Baseline or an infection requiring IV antibiotics within 4 weeks prior to Baseline
* Participant has active malignancy (except curatively resected squamous or basal cell carcinoma of the skin) requiring surgery, chemotherapy, or radiation within the prior 12 months (participants with a history of malignancy who have undergone curative resection or otherwise not requiring treatment for at least 12 months prior to Screening with no detectable recurrence are allowed).
* Participant has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has had suicidal ideation with at least some intent to act in the past 6 months as indicated by a positive response ("Yes") to either question 4 or question 5 of the "Screening/Baseline" version of the C-SSRS at Screening.
* Participant has alanine transaminase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >2.5x upper limit of normal (ULN)
* Participant has bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Participant has current unstable liver or biliary disease per Investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* QTc interval >450msec for male participants, QTc >470msec for female participants, or QTc >480 msec in participants with bundle branch block
* Participant has had recent surgery requiring general anesthesia within 2 weeks prior to Screening or is expected to have surgery requiring general anesthesia during the 12-week Main Treatment Period
* Participant has received a treatment with an experimental drug within 30 days or 5 half lives of the experimental drug (whichever is longer) prior to Baseline
* Participant has received treatment with rituximab within 6 months prior to Baseline or treatment is planned to occur during the study
* Participant has received treatment with intravenous immunoglobulin G (IVIG), SC immunoglobulin, or plasma exchange PLEX 4 weeks prior to Baseline or participant is on chronic IVIG, SC immunoglobulin, or PLEX
* Participant has previously participated in this study or participant has previously been assigned to treatment in a study of the medication under investigation in this study
* Participant has participated in another study of an investigational study medication (and/or an investigational device) within the previous 30 days or is currently participating in another study of an investigational study medication (and/or an investigational device)
* Participant has known positive serology for muscle-specific kinase

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (12):
- United States (12):
  - Mg0017 50564, Scottsdale, Arizona
  - Mg0017 50559, Los Angeles, California
  - Mg0017 50593, Rancho Mirage, California
  - Mg0017 50099, San Francisco, California
  - Mg0017 50557, O'Fallon, Illinois
  - Mg0017 50556, Chapel Hill, North Carolina
  - Mg0017 50086, Charlotte, North Carolina
  - Mg0017 50076, Columbus, Ohio
  - Mg0017 50555, Austin, Texas
  - Mg0017 50304, Dallas, Texas
  - Mg0017 50111, Seattle, Washington
  - Mg0017 50569, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Result] Freimer M, Desai U, Govindarajan R, Kang MK, Khan S, Khatri B, Levine T, Macwan S, Shieh PB, Weiss MD, Bloemers J, Boroojerdi B, Delicha EM, Lavrov A, Singh P, Howard JF Jr. Switching to subcutaneous zilucoplan from intravenous complement component 5 inhibitors in generalised myasthenia gravis: a phase IIIb, open-label study. Ther Adv Neurol Disord. 2025 Jul 5;18:17562864251347283. doi: 10.1177/17562864251347283. eCollection 2025. PMID 40620733

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in October 2022 and concluded in October 2024.
Pre-assignment Details: Participant Flow refers to the modified Intention to Treat Population (mITT).
Groups:
- Zilucoplan 0.3 mg/kg: Participants were administered zilucoplan (ZLP) 0.3 milligrams per kilogram per day (mg/kg/day) subcutaneously (SC) once daily (QD) for 12 weeks in Main Treatment Period. Participants who completed the 12-week Main Treatment Period without discontinuing study medication, continued to receive ZLP 0.3 mg/kg/day, SC, once daily in the Extension Treatment Period (up to approximately 84 weeks) until ZLP was commercially available or until further notice from the Sponsor.
Period: Main Treatment Period
Arm/Group | Zilucoplan 0.3 mg/kg
Started | 26
Completed | 23
Not Completed | 3
Not completed — Subject's lack of compliance with study procedures | 1
Not completed — Adverse Event | 2
Period: Extension Treatment Period
Arm/Group | Zilucoplan 0.3 mg/kg
Started | 23
Completed | 20
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the Modified Intention to Treat Population (mITT) which included all eligible study participants who received at least 1 post-baseline dose of study medication and had at least 1 post-Baseline assessment.
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (15.9)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 12
  65 - <85 years | 14
  >=85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 4
  White | 19
  Other or Mixed | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Over the Main Treatment Period
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE was defined as an AE starting on or after the time of first administration of investigational medicinal product (IMP) and up to and including 40 days after the final dose (or last contact depending on which occurs first).
Time Frame: From Baseline (Day 1) to Safety Follow-Up Visit (40 days post last dose) of Main Treatment Period (up to approximately 19 weeks)
Population: The Safety Set (SS) included all study participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
percentage of participants | 73.1

2. Primary Outcome: Percentage of Participants With TEAEs Leading to Withdrawal of Study Medication Over the Main Treatment Period
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE was defined as an AE starting on or after the time of first administration of IMP and up to and including 40 days after the final dose (or last contact depending on which occurs first).
Time Frame: as for outcome 1
Population: The SS included all study participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
percentage of participants | 7.7

3. Secondary Outcome: Change From Baseline to Week 12 in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Score
Description: The MG-ADL is a brief 8-item interviewer-administered patient-reported outcome (PRO) designed to evaluate MG symptom severity. The MG-ADL targets symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. Each item is assessed on a 4-point scale, where a score of 0 represents normal function and a score of 3 represents severely decreased ability to perform that function. The total MG-ADL score ranges from 0 to 24, with a higher score indicating more severe impairment. A positive change in score indicates worsening and negative change indicates improvement.
Time Frame: From Baseline to Week 12
Population: The modified ITT Population (mITT) population included all eligible study participants who received at least 1 post-Baseline dose of study medication and had at least 1 post-Baseline assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
score on a scale | -1.15 [-2.11 to -0.19]
Statistical Analysis 1: Comparison: Zilucoplan 0.3 mg/kg; Test type: Non-Inferiority — Non-inferiority of Week 12 MG-ADL over Baseline was shown if the upper limit of the 2-sided 95% confidence interval (CI) is less than 2; p < 0.001, Mixed Model for Repeated Measures (MMRM)

4. Secondary Outcome: Change From Baseline to Week 12 in the Quantitative Myasthenia Gravis (QMG) Score
Description: The QMG is a standardized and validated quantitative strength scoring system that included 13 items in the following categories: ocular and facial involvement, swallowing, speech, limb strength, and forced vital capacity. Scoring for each item ranges from no weakness (0) to severe weakness (3), with an overall score range from 0 to 39. Higher scores represent more severe impairment. A positive change in score indicates worsening and negative change indicates improvement.
Time Frame: From Baseline to Week 12
Population: The mITT population included all eligible study participants who received at least 1 post-Baseline dose of study medication and had at least 1 post-Baseline assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
score on a scale | -1.24 [-2.64 to 0.16]

5. Secondary Outcome: Percentage of Participants With Serious TEAEs Over the Main Treatment Period
Description: Treatment-emergent serious adverse events (serious TEAEs) were any untoward medical incidence in a participant during administered study treatment, whether or not these events were related to study treatment and additionally were emergent untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Required in patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent disability/incapacity
  * Was a congenital anomaly or birth defect
  * Important medical events
Time Frame: as for outcome 1
Population: The SS included all study participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
percentage of participants | 3.8

6. Secondary Outcome: Percentage of Participants With Study Withdrawal Over the Main Treatment Period
Description: Percentage of participants with study withdrawal based to pre-defined reasons in the protocol were reported.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 26
percentage of participants | 11.5

ADVERSE EVENTS:
Time Frame: From Baseline up to 84 weeks (Overall Treatment Period)
Description: A TEAE was defined as an adverse event (AE) starting on or after the time of first administration of IMP and up to and including 40 days after the final dose (or last contact depending on which occurs first). TEAEs were analyzed and reported for SS. The SS included all study participants who received at least 1 dose of study medication. The Overall Treatment Period is constituted of the Main Treatment Period and Extension Treatment Period.
Groups:
- Zilucoplan 0.3 mg/kg (Overall Treatment Period): Participants were administered zilucoplan (ZLP) 0.3 milligrams per kilogram per day (mg/kg/day) subcutaneously (SC) once daily (QD) for 12 weeks in Main Treatment Period. Participants who completed the 12-week Main Treatment Period without discontinuing study medication, continued to receive ZLP 0.3 mg/kg/day, SC, once daily in the Extension Treatment Period (up to approximately 84 weeks) until ZLP was commercially available or until further notice from the Sponsor.
Arm/Group | Zilucoplan 0.3 mg/kg (Overall Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 5/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilucoplan 0.3 mg/kg (Overall Treatment Period) (N=26)
Diverticulitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilucoplan 0.3 mg/kg (Overall Treatment Period) (N=26)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 2 (2)
Injection site pain (General disorders) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Amylase increased (Investigations) | 4 (6)
Lipase increased (Investigations) | 4 (5)
Injection site bruising (General disorders) | 2 (2)
Injection site pruritus (General disorders) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myasthenia gravis (Nervous system disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT05514873/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05514873/SAP_001.pdf